CLINICAL TRIAL: NCT05982509
Title: Clinical Trial to Assess the Efficacy and Safety of Neopop-S Containing EASYDEW
Brief Title: Clinical Trial to Assess the Efficacy and Safety of EASYDEW MD REGEN Cream Containing Neopop-S.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eun-ji Kim (Industry)
Responsible Party: Sponsor-Investigator, Eun-ji Kim, Clinical Trial Manager, CGBio Inc.
Organization: CGBio Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: G2204
Record Dates: First submitted 2023-07-28; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Laser-Induced Scar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention (No Intervention): Control group: 10 people without treatment
- Treatment (Experimental): Study Group: 10 People Applying EasyDew Regen MD Cream
  Interventions: Device: EasyDew Regen MD Cream

INTERVENTIONS:
Device: EasyDew Regen MD Cream — For the study group, I received the prescription Easy Dew Regen MD Cream from Picosure Laser Apply an appropriate amount twice a day (morning and evening) to the skin of the area so that it can be absorbed well do. The control group is the non-chalant group. However, for one month after the procedure, it is not a medical device The normal moisturizer you use at home is available, and the area where you have undergone laser treatment Apply it twice a day (morning and evening) to the skin so that it can be absorbed well.
  Arms: Treatment

SUMMARY:
The purpose of this clinical study is to evaluate the effect on skin regeneration after applying EasyDew MD Regen Cream containing Neopep-S, a regeneration factor, to patients who have undergone picosure picosure laser skin treatment as needed.

DETAILED DESCRIPTION:
This clinical study is a researcher-led randomized control group comparative clinical study that is conducted prospectively for one month after applying medical devices for clinical research.

The subjects are those who have undergone a picosure laser procedure for therapeutic purposes on the skin tissue of the face or body, and a screening test is conducted after the subject (and/or legal representative) agrees in writing to participate in the clinical study.

The screening test results are evaluated, and subjects who meet the selection criteria and do not meet the exclusion criteria are registered in clinical research.

Participating subjects are randomly assigned to the control group and the study group using a random number table at a 5:5 ratio.

* Control group: 10 people without treatment
* Study Group: 10 People Applying EasyDu Regen MD Cream Clinical study subjects are randomly assigned to control and study groups. In the case of the study group, the Easy Dew Regen MD cream provided through prescription is applied twice a day (morning and evening) to the skin of the area where the picosure laser treatment has been performed and absorbed well. The control group is the non-chalant group. However, general moisturizers that were used at home rather than medical devices for one month after the procedure can be used, and they are applied twice a day (morning and evening) to the skin of the area where the laser treatment has been performed and absorbed well.

One month of clinical research medical device application will be observed, and subjects will regularly visit the research institution to evaluate its validity and safety during screening visits (Visit1), treatment (Visit2), 2 weeks after treatment (Visit3), and 1 month after treatment (Visit3) You will receive it.

ELIGIBILITY:
Inclusion Criteria:

* Those aged 19 to 65 who have undergone picosure laser treatment on facial and body skin tissues
* Decided to participate in this clinical study and signed a written informed consent the subject

Exclusion Criteria:

* Subjects with uncontrolled diabetes
* Subjects with uncontrolled hypertension and cardiovascular disease
* Subjects with hemorrhagic diseases such as hemophilia
* Immunosuppressants, corticosteroids, cytotoxic agents, and anticoagulants can affect the results Subjects who are or are scheduled to receive medication for an extended period of time
* Acute or chronic skin disease causes stage progression or active bacteria in the application area Who has a virus infection
* When the researcher's judgment determines that participation in the study is inappropriate (e.g. keloid constitution)

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Transepidermal water loss Transcutaneous water loss (TEWL) measured | Before, immediately after treatment, and one month after application
  Before, immediately after treatment, and one month after application of the medical device Transcutaneous water loss (TEWL) measured

CONTACTS AND LOCATIONS:
Overall Officials: Jihye Lee, Study Director — CGBio Inc.
Locations (1):
- Ajou University Hospital, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim YH, Lee SJ, Kim HS, Woo SS, Kim MJ, Lim H, Lee IJ, Park YJ. Attenuation of Subclinical TNF-alpha Signalling in Xerotic Skin by AIMP-1 Derived Peptide Containing Moisturiser Leads to Skin Barrier Recovery. Exp Dermatol. 2025 Dec;34(12):e70183. doi: 10.1111/exd.70183. PMID 41355341